CLINICAL TRIAL: NCT00305149
Title: Use of Risk Factors for Initiation Therapy With Beacopp or Escalated Beacopp and Interim Evaluation and Modification of Therapy Based on Scintigraphy Results.
Brief Title: Risk Adapted Beacopp Regimen for Standard and High Risk Hodgkin Lymphoma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rambam Health Care Campus (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None
Other Study IDs: riskadapted beacopp/CTIL
Record Dates: First submitted 2006-03-20; First posted 2006-03-21 (Estimated); Last update posted 2006-03-21 (Estimated); Status verified 2006-03

CONDITIONS: Classical Hodgkin Lymphoma; Nodular Sclerosis; Mixed Cellularity; Lymphocyte Depletion; Lymphocyte Rich
Keywords: Hodgkin Lymphoma; BEACOPP; PET; Gallium; Tailored therapy
MeSH Terms: conditions — Hodgkin Disease

INTERVENTIONS:
Procedure: interim therapy scintigraphy study gallium scan or PET/CT
Procedure: "interim gallium or PET/CT"

SUMMARY:
.This study is trying to address change of chemotherapy dosage according to individual patient response to initial cycles of chemotherapy in order to reduce cumulative dose of chemotherapy.The study includes patients with early unfavorable and advanced hodgkin lymphoma. Patients with low risk were started with standard beacopp and only high risk patients were started with escalated beacopp.Following 2 cycles of therapy the patients were reassessed.Based on scintigraphy results decision was made regarding further therapylative chemotherapy for early responders and maximize dose intensity for late responders.

DETAILED DESCRIPTION:
Patients were eligible if they had early unfavorable disease or patients who presented with stage III or IV disease .Pt assigned to receive 6 cycles of Bleomycin Etoposide, Doxorubicin, Cyclophosphamide Procarbazine, Prednisone (BEACOPP) or increased dose BEACOPP. (IDB). Patient with Stage I or II with ³4 sites of disease, age ³50, ESR³50 "B" symptoms lymphocyte depleted histology "E" site, or bulky disease were defined as early unfavorable disease and were given standard BEACOPP (SB). Those with I, II B or bulky disease or Stage III, IV were defined according the IPS. Increased dose BEACOPP (IDB) cycles of therapy was initiated only to patients with IPS of 3 or more risk factors (high risk) Standard BEACOPP (SB) cycles were initiated to those with a score of 0-2 (standard risk). All patients had baseline GA67 or hybrid PET\CT scan at diagnosis and post first cycle for gallium scan or second cycle for hybrid PET\CT. Upon the scan results therapy was planned and given for addition of 4 cycles. Those with negative scan received cycles of SB as of the third cycle. Dose was reduced to level I to III if patient was hospitalized due to fever and neutropenia of 5 days or longer or pt had an episode of sepsis with unstable vital signs.

Patient with residual uptake interpreted as positive scan had additional cycles of IDB for a total of 6 cycles

ELIGIBILITY:
Inclusion Criteria:

* stage I-IIA/B with adverse prognostic or III-IV disease
* Age 18 and Over
* Performance status ECOG 0-3
* Hematopoietic WBC at least 4000/mm3(unless documented bone marrow involvement)
* Hepatic bilirubin no greater then 5 mg/dL
* RENAL:Creatinine no greater than 2.0mg/dL
* not pregnant or nursing
* Fertile patients must use effective contraception
* HIV negative
* No other malignancy within the past 5 years

Exclusion Criteria:

-

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130
Dates: Start 1999-07; Study Completion 2005-12

CONTACTS AND LOCATIONS:
Overall Officials: Ron Epelbaum, ND, Study Director — Rambam health care center, Bruce Rappaport Faculty of Medicine Technion
Locations (1):
- Eldad Dann, Haifa, Israel